CLINICAL TRIAL: NCT05018468
Title: Evaluation of the Quality of Ventilation With Facial Versus Nasal Mask After Induction of Anesthesia in Children 3 to 12 Years Old
Brief Title: Quality of Ventilation With Facial Versus Nasal Mask vs Nasal Mask Anesthesia in Children 3 to 12 Years Old
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Amir Shafa, Director, Isfahan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: IR.MUI.REC.1395.3.424
Record Dates: First submitted 2021-08-01; First posted 2021-08-24 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: Ventilation; Intubation Complication; Intubation; Difficult or Failed
MeSH Terms: conditions — Respiratory Aspiration | interventions — Masks

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ventilation with an anatomical facial mask (Experimental): Intervention group 1: Patients in this group undergo ventilation with an anatomical facial mask and 100% oxygen for three minutes. Intervention group 2: Patients in this group undergo ventilation with a nasal mask and 100% oxygen for three minutes. In both groups, ventilation will be performed with the controlled mode of the anesthesia machine with a volume of 8 cc/kg and a speed of 12-20/min.
  Interventions: Device: Ventilation
- ventilation with a nasal mask (Experimental): Intervention group 2: Patients in this group undergo ventilation with a nasal mask and 100% oxygen for three minutes. Ventilation will be performed with the controlled mode of the anesthesia machine with a volume of 8 cc/kg and a speed of 12-20/min.
  Interventions: Device: Ventilation

INTERVENTIONS:
Device: Ventilation — Patients in group 1 undergo ventilation with an anatomical facial mask and 100% oxygen for three minutes. Patients in group 2 undergo ventilation with a nasal mask and 100% oxygen for three minutes. In both groups, ventilation will be performed with the controlled mode of the anesthesia machine with a volume of 8 cc/kg and a speed of 12-20/min.
  Other Names: Mask

SUMMARY:
In this single-blind clinical trial study, 70children who are candidates for lower abdominal elective surgery under general anesthesia presented at Imam Hossein Hospital in Isfahan will be included in the study and will be divided into 2 groups. In the first group, ventilation with facial mask and in the second group, ventilation with nasal mask will be done for three minutes. Then the reduction in SPO2 and the impossibility of ventilation of patients will be evaluated and compared between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Age category between 3 to 12 years
* Candidate for lower abdominal elective surgery under general anesthesia
* No obstruction in the nasal pathway
* No deformity and fractures in facial
* No acute or chronic lung disease

Exclusion Criteria:

* Impossibility of airway oropharyngeal ventilation
* Impossibility of ventilation of the anatomical facial mask with neck extension
* Dissatisfaction with participating in the study.

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-06-20 (Actual)

PRIMARY OUTCOMES:
Average airway pressure | change from baseline at five minutes after incubation
  Ventilation device
Average End-tidal CO2 (EtCO2) | change from baseline at five minutes after incubation
  Ventilation device
Average Oxygen saturation (SpO2) | change from baseline at five minutes after incubation
  Ventilation device

CONTACTS AND LOCATIONS:
Locations (1):
- Alzahra Hospital, Isfahan, Iran

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol